CLINICAL TRIAL: NCT05234463
Title: Study of the Link Between Complement Activation and IgA Nephropathy Severity
Acronym: ICONE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8361
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: IgA Nephropathy Severity in Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples (14mL) in dry tubes for isolation of serum
  * EDTA-blood (4,5mL) for EDTA plasma and DNA extraction
  * Citrated plasma (9mL)
  * Urine (10mL)
  * Paraffin-embedded and frozen kidney or graft biopsy specimen for complement immunomarquage (residues of biopsies realized in clinical practice, on a selected subset of patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IgAN patients — Adult patients Histologically proven diagnosis of IgA nephropathy Primary and secondary forms of the disease With or without kidney transplantation history Regardless of kidney/graft function Patients followed in the Nephrology Department of Strasbourg University Hospital.

SUMMARY:
ICONE study (IgA Complement and NEphropathy is a prospective monocentric observational study.

The main objective is to evaluate the relevance of complement activation as a biomarker of disease severity and progression in patients with a biopsy proven IgAN.

DETAILED DESCRIPTION:
IgA nephropathy (IgAN) is a common cause of glomerulonephritis and a major cause of end stage renal disease in up to 20-40% of patients. However, its prognosis still cannot be accurately predicted due to the high heterogenicity of clinical presentations and courses. Complement dysregulation is a main driver of glomerular damages in many glomerulonephritis. Given the growing body of evidence of complement lectin/alternative pathways activation in IgAN pathogenesis, the investigators propose the evaluation of a combination of biomarkers of infra-clinical complement activation to stratify the risk of disease's progression. This study aims to identify subsets of patients in whom complement activation plays a critical role in disease progression. This is of particular interest in the aera of emergence of complement-targeting therapies in IgAN

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, male or female, with a biopsy proven IgA nephropathy.
* Primitive and secondary forms can be included
* Regardless of the date of diagnosis and the level of kidney function
* With or without past of kidney transplantation
* Followed in the Nephrology Department, Strasbourg University Hospital
* Signed informed consent

Exclusion Criteria:

* Active or recent infectious or inflammatory syndrome (<2 months), recent vaccination (<2 months), ongoing acute humoral rejection treatment, treatment with plasma exchanges (<2 months), current treatment with complement inhibitors
* Impossibility of giving informed information (emergency situation, difficulties in understanding, etc.)
* Subject under safeguard of justice, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a histologically proven diagnosis of IgA nephropathy, with or without kidney transplantation history followed in the Nephrology Department of Strasbourg University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of a severe form of IgA nephropathy | At inclusion
  Occurrence of a severe form of IgA nephropathy, with at least one of the following severity criteria: i) a rapid decline in estimated glomerular filtration rate the incidence of end stage kidney disease, iii) the presence of malignant hypertension or thrombotic microangiopathy features, iv) histological endo and/or extra capillary proliferation (E1 and/or C1 according to Oxford 2016 MEST-C score).
  Infra-clinical complement activation is defined as a sC5b-9 > 300ng/mL in plasma or a positive ex vivo complement activation functional test on endothelial cells.
Incidence of a severe form of IgA nephropathy | 1 year after inclusion
  Occurrence of a severe form of IgA nephropathy, with at least one of the following severity criteria: i) a rapid decline in estimated glomerular filtration rate the presence of malignant hypertension or thrombotic microangiopathy features, iv) histological endo and/or extra capillary proliferation (E1 and/or C1 according to Oxford 2016 MEST-C score).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de néphrologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No